CLINICAL TRIAL: NCT07362602
Title: Exploratory Study on in Vivo CAR-T Therapy Targeting CD20 for the Treatment of Hematological Malignancies
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army (Other)
Responsible Party: Principal Investigator, Xiaolin Yin, Professor, The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CD20-IIT-B cell malignancies
Record Dates: First submitted 2026-01-05; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in vivo CAR-T drug, Escalation doses (Experimental): In vivo CAR-T drug targeting CD20 based on mRNA-LNP
  Interventions: Drug: In vivo CAR-T drug targeting CD20 based on mRNA-LNP
- in vivo CAR-T drug, Extended doses (Experimental): In vivo CAR-T drug targeting CD20 based on mRNA-LNP
  Interventions: Drug: In vivo CAR-T drug targeting CD20 based on mRNA-LNP

INTERVENTIONS:
Drug: In vivo CAR-T drug targeting CD20 based on mRNA-LNP — In vivo CAR-T drug targeting CD20 based on mRNA-LNP

SUMMARY:
Malignant hematological tumors mainly derived from adult B cells are mainly acute lymphoblastic leukemia (ALL) and non Hodgkin lymphoma (NHL). Overall, although existing therapies have significantly improved the survival rates of most patients, the treatment of relapsed/refractory patients still faces significant challenges. CD20 is a transmembrane protein highly expressed on the surface of B cells, almost penetrating the precursor, mature, and activated stages of B cells, but lacking in plasma cells, making it an ideal target for B cell malignancies.

In recent years, the breakthrough development of in vivo CAR-T therapy has overturned the traditional paradigm of in vitro CAR-T technology. The core principle is to directly deliver the gene encoding chimeric antigen receptor (CAR) to T cells in the patient's body through gene delivery vectors, without the need for in vitro isolation, modification, and amplification processes, and to complete the gene reprogramming of T cells in vivo. At present, the mainstream carrier technologies for CAR-T therapy in vivo are divided into two categories: lentiviral carriers and lipid nanoparticle (LNP) carriers. LNP carriers have significantly broken through the clinical bottlenecks of traditional CAR-T in terms of cost and accessibility, safety, and timeliness.

This experimental drug is a CD20 based messenger ribonucleic acid (mRNA) therapeutic drug, which is an injection formed by loading mRNA onto lipid nanoparticles (LNP). It has shown efficient B-cell clearance activity and good safety in non clinical settings, supporting further clinical exploration in B-cell hematological malignancies. It is expected to provide an innovative, safe, and accessible immunotherapy for B-cell hematological malignancies and bring better clinical benefits to more patients with B-cell hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range of 18-70 years old, gender not limited;
* 2. Expected survival time exceeds 12 weeks;
* 3. Diagnosed with blood system tumors such as CD20+B-cell lymphoma or lymphocytic leukemia and meeting the corresponding previous treatment requirements;
* 4. There are assessable lesions (applicable only to lymphoma patients);
* 5. The physical fitness status score of the Eastern Cancer Collaboration Group (ECOG) is 0 or 1 point; Before screening (at baseline), corresponding requirements should be met;
* 7. Male and female patients of appropriate age must use reliable methods of contraception before entering the trial, during the research process until 30 days after discontinuation of medication; Reliable contraceptive methods will be determined by the primary researchers or designated personnel;
* 8. Those who can understand this experiment and have signed the informed consent form.

Exclusion Criteria:

* 1. Accompanied by other uncontrolled malignant tumors;
* 2. Received chimeric antigen receptor therapy or other transgenic T cell therapy within 6 months;
* 3. Known history of HIV or hepatitis B (HBsAg positive and HBV DNA reaching the detection limit) or hepatitis C virus (anti HCV positive) infection;
* 4. Participants with a history of CNS lymphoma, malignant cells in cerebrospinal fluid, or brain metastases;
* 5. Participants with atrial or ventricular involvement;
* 6. Emergency treatment is required due to the impact of tumor masses, such as intestinal obstruction or vascular compression;
* 7. Suffering from serious diseases such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis, cerebral hemorrhage, poorly controlled hypertension, or other uncontrolled active diseases that hinder participation in the trial;
* 8. Unstable pulmonary embolism, deep vein thrombosis, or other major arterial/venous thromboembolism events occurred within 30 days prior to enrollment. If receiving anticoagulant therapy, the treatment dose of participants must reach a stable level before enrollment;
* 9. For those who have been using immunosuppressants for a long time after organ transplantation, except for recent or current inhaled corticosteroid therapy;
* 10. Any pregnant or breastfeeding woman, or participant who plans to conceive during or within 18 months after treatment;
* 11. Within 14 days prior to enrollment, there is an active or uncontrollable infection that requires systemic treatment (excluding simple urinary tract infections or upper respiratory tract infections).
* 12. The researcher believes that there are any other factors that are not suitable for the study participants to enter this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Within 28 days after the initial treatment
The incidence of adverse effects | Through study completion, an average of 2 years
Maximum tolerated dose (MTD) or optimal biological dose (OBD) | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
0bjective response rate (ORR) | Through study completion, an average of 2 years
Disease control rate (DCR) | Through study completion, an average of 2 years
Duration of response (DoR) | From the date of the first PR/CR to the date of first comfired progression or date of death from any cause, whichever came first, assessed up to 24 months
Progression free survival (PFS) | From date of initial treatment until the date of first comfired progression or date of death from any cause, whichever came first, assessed up to 24 months